CLINICAL TRIAL: NCT00248196
Title: COOL MI II: Cooling as an Adjunctive Therapy to Percutaneous Intervention in Patients With Acute Myocardial Infarction
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radiant Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50-0045
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2007-08

CONDITIONS: Acute Myocardial Infarction

INTERVENTIONS:
Device: Reprieve Endovascular Temperature Therapy System

SUMMARY:
Coronary heart disease is the single leading cause of death in the United States. In 2000, it was implicated in 681,000 deaths (1 in every 5 deaths). Myocardial infarction (MI) is the major cause of death in patients dying of coronary heart disease, with an estimated incidence of 1.1 million new and recurrent cases per year. It is well established that reperfusion is the most successful treatment for salvaging myocardium during acute infarction. However, despite such treatment, a substantial number of patients still remain at risk of developing large infarcts, with reduced left ventricular function and increased mortality. Therefore, adjunctive therapies that are designed to reduce ischemic metabolism and cellular injury pending successful reperfusion, or to protect myocytes against the undesired effects of reperfusion ("reperfusion injury"), should be beneficial in limiting infarct size. Mild hypothermia is one such potential therapy. This study has been designed to evaluate whether the adjunctive use of mild hypothermia further reduces the extent of heart damage caused by a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* The patient is greater than 18 years of age.
* The patient must have symptoms consistent with acute myocardial infarction (i.e. chest pain, arm pain, etc.) and unresponsive to nitroglycerin, with symptoms beginning greater than 30 minutes but less than 6 hours prior to presentation.
* Anterior wall MI with ST-segment elevation of ≥ 1 mm in two or more contiguous leads.
* The patient is eligible for percutaneous coronary intervention (PCI).
* The expected timing of the treatment pathway for the patient will allow for at least 30 minutes of cooling prior to PCI.
* The patient or patient legal guardian is willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* The patient has had a previous myocardial infarction within one month.
* The patient is experiencing cardiogenic shock (systolic blood pressure [SBP] <80 mmHg and non-responsive to fluids, or SBP <100 mmHg with vasopressors, or requirement for an intra-aortic balloon pump [IABP]).
* The patient has a known hypersensitivity to hypothermia, including a history of Raynaud's disease.
* The patient has a known hypersensitivity or contraindication to aspirin, heparin, or sensitivity to contrast media, which cannot be adequately pre-medicated.
* The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia or sickle cell anemia, or will refuse blood transfusions.
* The patient has a height of <1.5 m (4 feet 11 inches).
* The patient is known to be pregnant or is expected to become pregnant prior to the 1 month follow-up.
* The patient has a known hypersensitivity to buspirone hydrochloride or meperidine and/or has been treated with a monoamine oxidase inhibitor in the past 14 days.
* Patient has a known history of severe hepatic or renal impairment, untreated hypothyroidism, Addison's disease, benign prostatic hypertrophy, or urethral stricture, that in the opinion of the physician would be incompatible with meperidine administration.
* The patient has an inferior vena cava filter in place.
* The patient has a pre-MI life expectancy of <1 year due to underlying medical conditions or pre-existing co-morbidities.
* The patient has a known, unresolved history of drug use or alcohol dependency, or lacks the ability to comprehend or follow instructions.
* The patient is currently enrolled in the COOL MI trial or in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with the COOL MI study endpoints. Note: For the purpose of this protocol, patients involved in extended follow-up trials for products that were investigational but are currently commercially available are not considered enrolled in an investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2005-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Reduction in infarct size (single photon emission computed tomography [SPECT])
Equivalent safety profile

SECONDARY OUTCOMES:
Reduction in infarct size (creatinine kinase MB [CK-MB], ST- Segment Resolution)
Improvement in left ventricular ejection fraction (LVEF)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Carrozza, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Simon R Dixon, MBChB, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan